CLINICAL TRIAL: NCT01887925
Title: The Effects of Per3, Clock Polymorphism on Sleep and Associated Symptoms in Breast Cancer Patients Under Chemotherapy.
Brief Title: The Effects of Circadian Gene on Sleep and Associated Symptoms in Breast Cancer Patients Under Chemotherapy
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bong-Jin Hahm, professor, Seoul National University Hospital
Other Study IDs: BreastCaCTx_circadian
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; sleep; anxiety; depression; life quality
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- breast cancer: breast cancer patients receiving chemotherapy

SUMMARY:
The purpose of this study is the evaluation of effect of circadian gene on sleep and other symptoms in breast cancer patients under chemotherapy.

DETAILED DESCRIPTION:
In this study, the investigators are going to examine the effect of genetic polymorphism on sleep, anxiety, depression and other cancer-related symptoms in patients with breast cancer who have started chemotherapy after surgery. No intervention was intended and blood sample was taken with other routine laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* Patient with breast cancer without metastasis
* Patient received cancer surgery and medically stable
* Patient will undergo chemotherapy for the first time in life
* Patient have signed on the informed consent, and well understood the objective and procedure of this study

Exclusion Criteria:

* Patient received chemotherapy or radiotherapy
* Patient had another cancer before
* Patient have metastasis
* Patient with severe medical condition
* Patient had taken psychiatric medication more than 1 month in life
* Patient worked the night shift for more than 1 month in 6 months

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: university hospital, oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Sleep Impairment at 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Sleep impairment will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.

SECONDARY OUTCOMES:
Changes from Baseline Quality of Life at 1 Month After Chemotherapy | baseline, 1 month after chemotherpy completion
  Quality of life will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month after completion of the chemotherapy.
Changes from Baseline Cancer-related Symptoms at 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Cancer-related symptoms will be evaluated by questionnaires before chemotherapy.
  The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.
Changes from Baseline Fatigue at 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Fatigue will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.
Changes from Baseline Depression at 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Depression will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.
Changes from Baseline Anxiety 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Anxiety will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.
Changes from Baseline PTSD Symptoms 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  PTSD symptoms will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.
Changes from Baseline Menopausal Symptoms 1 Month After Chemotherapy | baseline, 1 month, 3 months, 1 month after chemotherpy completion
  Menopausal symptoms will be evaluated by questionnaires before chemotherapy. The evaluation will be followed 1 month, 3 months after starting chemotherapy. The final evaluation will be done 1 month after completion of the chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Jin Hahm, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- [Derived] Son KL, Jung D, Lee KM, Yeom CW, Oh GH, Kim TY, Im SA, Lee KH, Spiegel D, Hahm BJ. Morning Chronotype Decreases the Risk of Chemotherapy-Induced Peripheral Neuropathy in Women With Breast Cancer. J Korean Med Sci. 2022 Feb 7;37(5):e34. doi: 10.3346/jkms.2022.37.e34. PMID 35132840
- See also: study site — http://www.snuh.org/